CLINICAL TRIAL: NCT01029561
Title: Impact of Obstructive Sleep Apnea Syndrome on Metabolic Syndrome in Severe Obesity
Acronym: SYBILA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); August Pi Sunyer Biomedical Research Institute (Other)
Responsible Party: Carmen Monasterio i Ponsa, Institut d'Investigació Biomèdica de Bellvitge(IDIBELL)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI08/0800; Beca SEPAR. Num. Ref: 736 (Other Grant/Funding Number: SPANISH RESPIRATORY SOCIETY: 736)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 2009-10

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Adipokines; Cytokines
Keywords: Metabolic syndrome; Insulin Resistance; Adipokines; Proinflammatory markers; Obstructive Sleep Apnea Syndrome; Continuous Positive Airway Pressure; Obesity; Bariatric surgery
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Sleep Apnea, Obstructive; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP and diet (Active Comparator): The patients with severe OSA (AHI>=30) who do not fulfill the specific exclusion criteria wil be randomized. In the CPAP and diet arm, patients wil receive Continuous Positive air pressure therapy and the regular dietary treatment.
  Interventions: Device: CPAP; Behavioral: Diet
- Diet (Active Comparator): The diet arm wil receive the Conventional diet treatment that usually receive the patients included in the Bariatric Surgery Program
  Interventions: Behavioral: Diet

INTERVENTIONS:
Device: CPAP — Treatment with Continuous Positive Airway Pressure
  Arms: CPAP and diet
Behavioral: Diet — Conventional diet treatment that undergo patients in the Bariatric Surgery Program

SUMMARY:
The aim of this project is to study the relationship between obstructive sleep apnea (OSA) and metabolic syndrome (MS) in a population of obese patients who are candidates for bariatric surgery. The investigators will study the influence of OSA through hypoxia and sleep fragmentation on different proinflammatory adipokines and cytokines, on metabolic syndrome and on insulin resistance, as well as how these respond to treatment with continuous positive airway pressure (CPAP).

In the first part of the study (part A) the investigators will perform an observational study of cases and controls. Based on the diagnostic polysomnography the patients will be divided into two groups depending on their apnea-hypopnea index (AHI): OSA (AHI >= 15/h) and non-OSA (AHI <15/h). The results will be analyzed depending on the presence or not of OSA.

In the second part of the study (part B), the patients with severe OSA (AHI ≥ 30/h) will be randomized into two groups: one group will receive CPAP + diet treatment and the other group will only receive diet treatment. After 3 months of treatment (CPAP + diet vs. diet), the investigators will analyze the overall effect on metabolic syndrome and the effect on its individual components, as well as the above-mentioned inflammatory pathways and insulin sensitivity, between the 2 groups. This will be carried out through a randomized controlled study in which the investigators will compare the effect of CPAP with the effect of conservative treatment.

DETAILED DESCRIPTION:
METHODOLOGY

PARTICIPATING CENTERS: Respiratory Medicine and Endocrinology Services of the Hospital Universitari de Bellvitge, of the Hospital de la Santa Creu i Sant Pau and of Hospital Clínic de Barcelona.

PATIENTS (recorded in eligibility criteria)

Ethical aspects: All patients will be asked for informed consent in accordance with the procedures of the Ethical Committee of the hospitals. Patients will be recruited in the initial stage of the protocol and waiting list for bariatric surgery. Currently the waiting list is 2 to 3 years long and the patients are screened for OSA in the year before the intervention, with the aim of treating OSA patients in order to reduce the perioperative surgical risk. Therefore the protocol will not lead to a delay in the start of treatment, since treatment will be commenced earlier than usual. Once the study period is over, the patients in the control group will receive CPAP if necessary.

DESIGN:

Multi-center study (with the participation of 3 centers), with an initial part (A) that is an observational prospective case-control study coordinated by the Hospital Universitari de Bellvitge. Based on the polysomnography performed on all patients who fulfill the inclusion criteria, the patients will be put into two groups: CASES: patients with OSA (AHI >= 15) and CONTROLS: Non-OSA (AHI < 15). We will analyze whether metabolic syndrome is present or not and the different determinations depending on whether or not the patients have OSA. In the second part of the study (B) coordinated by the Hospital de la Santa Creu i Sant Pau we will analyze the treatment response of OSA patients with AHI >= 30 to CPAP with a prospective, controlled and randomized study of parallel groups, in which CPAP treatment will be compared with conservative treatment in the form of a diet.

Sample Size:

In the observational study (part A), based on previous studies and accepting an alpha risk of 0.05 and a beta risk of 0.20 in bilateral contrast, we calculated that 39 subjects are needed in each group to detect a difference greater than or equal to 0.32 between them. A proportion of 0.55 is assumed in one of the groups. The dropout rate for the study has been estimated at 10%. The ARCCOSINE approximation has been used.

In the treatment response study (part B), 63 subjects are needed in each group to detect a difference that is greater or equal to 1 units of HOMA, assuming a standard deviation of 1.90 based on previous studies. The dropout rate for the study has been estimated at 10%.

STUDY VARIABLES:

1. Anthropometric and demographic data: age, sex, weight, height, BMI, neck circumference. Time between when patient became obese and recruitment date (period of obesity).
2. Measures of central obesity: waist circumference (above the superior border of the iliac crest). The body mass index will be determined by dividing the weight in kilograms by the height in meters squared. The waist/hip ratio will be measured.
3. Body fat composition will be measured with electrical bioimpedance using the Bioimpedance Meter BIA 101 (Akern Bioresearch, Florence, Italy), with an analyzer for bioimpedance of the vectors R (resistance) and Xc (reactance) with reference values for obese subjects (Piccoli A. et al. Int. Journ. Of Obesity 1998; 22:97-104).
4. General clinical questionnaire: cardiovascular risk factors and co-morbidity.
5. Self-assessment of daytime sleepiness. This will be analyzed using the Epworth scale (MW Johns, Sleep 1991, 14;540).
6. Degree of sleepiness according to the definition of the American Thoracic Society: classification into three categories: light, moderate and severe somnolence.
7. Hours of sleep: this will be analyzed using a sleep diary that will be kept during a period of 15 consecutive days. In addition, basic questions will be asked of each patient while obtaining the medical history about the usual hours of sleep on working days and weekends and holidays.
8. Physical activity questionnaire: international self-administered questionnaire of physical activity, short version. International physical activity questionnaire (IPAQ) www.ipaq.ki.se.
9. Questionnaire on quality of life in patients with sleep apnea Quebec Sleep Questionnaire (QSQ), self-administered, version translated into Spanish. (Y Lacasse, Thorax 2004).
10. Respiratory Function Study: maximum F/V loop performed with Datospir 500 spirometer (SIBEL, Barcelona), in accordance with the norms and reference values of the SEPAR (Roca et al. Bull Eur Physiopathol Respir, 1986, 22: 217-24). In addition to the spirometric variables (FVC; FEV1, FEV1/FVC,PEF), MIF50, MEF50/MIF50, PEF/FEV1 FEV0,5/FEV1, VVM/FEV1 will also be assessed. Static lung volumes. Helium dilution technique in accordance with the norms and reference values of the SEPAR (Roca el al. Bull Eur Physiopathology Respir, 1986, 22: 217-224). Arterial gases will be taken at rest while the subject is seated and breathing room air and they will be evaluated using the established recommendations (SEPAR working group for the practice of arterial gasometry (Arch. Bronconeumol 1998: 34: 142-151).
11. Conventional Polysomnography (PSG). This will be performed over an entire night using a Compumedics Siesta Polysomnograph (Compumedics, Melbourne, Australia). It will include 2 electroencephalogram channels, 2 electro-oculography channels, chin electromyography, oronasal flow measured by a thermistor and nasal canula, thoracic and abdominal excursion bands, oxyhaemoglobin saturation (SpO2) measured with a finger probe, electrocardiogram, anterior tibial electromyogram, sound recording for snores, and a body position sensor. The criteria of Rechtstaffen and Kales will be used for visual scoring of sleep stages. The minimum recording time is 6 hours and the minimum sleep time is 3 hours. Definition of apnea: absence of flow for at least 10 seconds. Definition of hypopnea: any reduction of flow with a minimum duration of at least 10 seconds that is accompanied by a desaturation (greater or equal to 3%) and/or a transitory awakening or arousal (with arousal defined according to ASDA criteria: Sleep, 1992; 15: 173-184). Definition of hypoventilation: prolonged periods of arterial desaturation not preceded by episodes of respiratory events. The following data will be recorded: number of apnea/hypopnea episodes per hour (AHI), percentage of time in apnea and/or hypopnea, number of arousals/hour, sleep efficiency (total sleep time/length of recording), percentage of time in phases 1, 2, 3-4 and REM, initial oxyhemoglobin saturation, average of oxyhemoglobin saturation, minimum saturation, time with saturation of oxyhemoblobin under 90 % (CT90) and 85 % (CT85).
12. Blood tests: a blood sample will be taken from all patients to determine their biochemical profile and full general blood count, lipid profile (Triglycerides, cholesterol (total cholesterol, HDL, VDL, LDL), glycosylated hemoglobin, insulin, leptin, TNF alpha, TNF alpha soluble receptors 1 and 2, IL-6, IL-8 and adiponectin.
13. Measurement of blood pressure: The morning after the PSG is carried out 2 blood pressure measurements will be taken at rest in a supine position, separated by 5 minutes, and additional measurements will be made if there is a difference of more than 5 mmHg between them. In accordance with the rules of the Sociedad Española de Hipertensión. (Hipertension 2005; 22 supl 2: 16-20)
14. Calculation of insulin resistance: This will be performed using the HOMA calculation (Homeostasis Model Assessment) modeled by Matthews et al (Diabetologia 1985; 28: 412-419.).
15. Glucose tolerance measurements: In those patients without recognized diabetes mellitus, a glucose load will be given after 12 hours of fasting, by administering 75 g of glucose and determining glucose levels at 0 and 120 minutes.
16. Metabolic Syndrome: The percentage of Metabolic Syndrome will be defined for each of the groups, with Metabolic Syndrome defined in accordance with international criteria (Adult Treatment Panel III. JAMA 2001; 2486-2497) as the existence of the following three conditions: 1) Central obesity: waist > 88 cm in women, > 102 cm in men, 2) Arterial hypertension: AHT greater than or equal to 130/85 mmHg or treatment, 3) Hyperglycemia: plasma glucose > 6.1 mmol/L, 4) Hypertriglyceridemia: TG greater than 1.7 mmol/L, 5) Hypo-HDL: HDL less than 1.3 mmol/L in men and 1 mmol/L in women. A metabolic index will be established for each subject that will define the number of individual components of Metabolic Syndrome they present.

PROCEDURE:

Part A: All patients from the obesity surgery program of the Endocrinology service that fulfill the inclusion criteria will be recruited. Patients will be assigned to groups according to the result of the polysomnography. Patients with AHI >= 15 will be considered OSA and all other patients non-OSA until there are 39 patients in each group, in accordance with the sample calculation. Thus all patients will be evaluated at baseline according to their condition of OSA/non-OSA.

Part B: Subsequently, the patients with severe OSA (AHI>=30) who do not fulfill the specific exclusion criteria for part B will randomized into the group for treatment with CPAP and diet or the group for conservative treatment (diet). The patients will be evaluated after 6 and 12 weeks from the start of treatment (CPAP and diet vs. diet). The variables will be determined at baseline and after 12 weeks.

STATISTICAL ANALYSIS:

A descriptive analysis of the sample will be carried out in accordance with central tendency measures (mean, median) and dispersion measures (standard deviation and interquartile range) in accordance with normality criteria (Kolmogorov-Smirnov test). Then a comparative study will be performed between the groups using chi-square test or Fisher's exact test as appropriate to the qualitative variables; and Student's t test or the Mann-Whitney U test will be used for the quantitative variables according to normality criteria.

The percentages of metabolic syndrome in the OSA and non-OSA patients, as well as the percentages of OSA in the groups with and without metabolic syndrome will be compared. The differences in metabolic syndrome and the metabolic index will be analyzed according to the severity of the OSA. This will initially be carried out through the univariate analysis of the variables gathered in the group of patients and the control groups, and those variables that have an association with p-value < 0.10, and that do not interact among themselves will be considered in a binary logistic regression model.

In the second part of the study, after 12 weeks of CPAP treatment, the variables from the baseline and final situation will be compared with the parametric or non-parametric tests as appropriate depending on their normality.

The analysis will be carried out using the statistical package SPSS 15.0 (Illinois, Chicago), and a p-value < 0.05 will be considered statistically significant in all cases.

ELIGIBILITY:
Inclusion Criteria for part A:

Patients who are included in the obesity surgery program will be recruited if they fulfill the following criteria:

* Age between 18 and 65 years.
* Body mass index (BMI) >40 kg/m2 or BMI > 35 kg/m2 with co-morbidity related to obesity.

Inclusion Criteria for part B:

In the treatment response study we will include patients diagnosed at the baseline polysomnography with severe OSA (AHI >= 30) who fulfill the inclusion criteria for part A and who do not present specific exclusion criteria for part B.

General Exclusion Criteria (for part A):

* Prior treatment with CPAP.
* Severe or unstable cardiovascular disease (severe or surgically treated valvulopathy, myocardial infarction, unstable angina, cardiac surgery) during the 6 months prior to inclusion in the study.
* Evidence of acute or chronic inflammatory illness different to obesity itself (connective tissue disease, active neoplasia) or associated infectious process during the 6 weeks prior to inclusion in the study.
* Severe cognitive or psychiatric disorder that would make it difficult to complete the clinical questionnaires.
* Severe chronic diseases that may interfere in a significant way with the results of the study.
* Chronic obstructive pulmonary disease defined by FEV1/FVC < 0.7.
* Pregnancy.
* Alcohol abuse (daily alcohol consumption >80 g).
* Express decision of the patient to not participate in the study.

Exclusion Criteria for part B:

* Severe or incapacitating somnolence.
* Professional drivers or users of dangerous machinery.
* Congestive cardiac insufficiency or significant valvulopathy or chronic cor pulmonale.
* Use of oral anti-diabetic drugs or insulin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-06 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
To analyze the effect of CPAP treatment on insulin resistance and metabolic syndrome in patients with severe obesity and OSA. | baseline and after 12 weeks of CPAP

SECONDARY OUTCOMES:
To study the relationship between OSA and metabolic syndrome in a population of severely obese patients who are candidates for bariatric surgery. | baseline and after 12 weeks of CPAP
To study the influence of OSA on proinflammatory markers and on different adipokines in severely obese patients and their relationship with metabolic syndrome, insulin resistance and body composition. | baseline and after 12 weeks of CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Monasterio, MD, Principal Investigator — Institut d´Investigació de Bellvitge (IDIBELL)
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Barcelo A, Morell-Garcia D, Salord N, Esquinas C, Perez G, Perez A, Monasterio C, Gasa M, Fortuna AM, Montserrat JM, Mayos M. A randomized controlled trial: branched-chain amino acid levels and glucose metabolism in patients with obesity and sleep apnea. J Sleep Res. 2017 Dec;26(6):773-781. doi: 10.1111/jsr.12551. Epub 2017 May 17. PMID 28513068
- [Derived] Salord N, Fortuna AM, Monasterio C, Gasa M, Perez A, Bonsignore MR, Vilarrasa N, Montserrat JM, Mayos M. A Randomized Controlled Trial of Continuous Positive Airway Pressure on Glucose Tolerance in Obese Patients with Obstructive Sleep Apnea. Sleep. 2016 Jan 1;39(1):35-41. doi: 10.5665/sleep.5312. PMID 26350474